CLINICAL TRIAL: NCT00592748
Title: Randomized Study of Charged Particle RT for Chordomas and Chondrosarcomas of the Base of Skull or Cervical Spine
Brief Title: Charged Particle RT for Chordomas and Chondrosarcomas of the Base of Skull or Cervical Spine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Norbert J. Liebsch, M.D., Director, Skull-Based Service, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97-553
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Chordoma; Chondrosarcoma
Keywords: charged particle radiation therapy
MeSH Terms: conditions — Chordoma; Chondrosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): 40-44 Treatments
  Interventions: Radiation: Charged Particle Radiation Therapy
- Group 2 (Active Comparator): 37-40 Treatments
  Interventions: Radiation: Charged Particle Radiation Therapy

INTERVENTIONS:
Radiation: Charged Particle Radiation Therapy — Radiation doses will be determined by planning CT

SUMMARY:
The primary purpose of this study is to determine if the administration of a higher dose would decrease the chance of tumor recurrence, compared to the risk of tumor recurrence with a lower dose. Most of the treatment will be given protons, but participants may receive a small portion of treatment with x-rays, because less radiation is given to the skin with x-rays. This study uses two slightly different doses of radiation It is not clear at this time which of the dose levels is better.

DETAILED DESCRIPTION:
* Participants will be assigned to a dose level by random chance, like flipping a coin.
* A treatment plan will be determined by a treatment planning CT scan and will either involve 40-44 treatments or 37-40 treatments.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven chordoma. Slides must be reviewed prior to randomization by the central review pathologist
* Sites: Intercranial (sphenoid, clivus, petrous, basio-occiput) or cervical spine
* Boost target volume less than or equal to 150
* 18 years of age or older
* Karnofsky Performance Status > 50
* Neurologic Function of I or II
* No evidence of metastases

Exclusion Criteria:

* Previous radiation to the head or neck that would compromise the ability to deliver the prescribed treatment
* Concurrent or prior malignancy unless disease free for 5 or more years
* Evidence of metastatic disease
* Diabetes mellitus
* Major medical illness or psychiatric impairments that in the opinion of the investigator, will prevent administration or completion of the protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 1999-06; Primary Completion 2007-07 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Acute Toxicity | 90 days

SECONDARY OUTCOMES:
Establish local control rates for both dose schedules. | 5 years
To provide date to be used as the basis for choosing the dose of charged particle radiation for chordomas of the base of skull and the cervical spine. | 5 years
Late Toxicity | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Norbert J. Liebsch, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States